CLINICAL TRIAL: NCT04277156
Title: A Two-strain Probiotic (L Rhamnosus ATCC 53103 & L Reuteri DSM 29063) Compared With a Single Strain Probiotic (L Rhamnosus ATCC 53103) for Preventing Antibiotic-associated Diarrhea: an Open-label, Randomized, Noninferiority Trial
Brief Title: L Rhamnosus ATCC 53103 & L Reuteri DSM 29063 Compared With L Rhamnosus ATCC 53103 for Preventing AAD in Children
Acronym: FLOSTRUM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Adamed Pharma S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FLOSTRUM2020
Record Dates: First submitted 2020-02-10; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-01

CONDITIONS: Antibiotic-associated Diarrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flostrum Baby (Experimental): The test product will be Flostrum Baby, which is a food supplement consisting of two bacterial strains: Lactobacillus rhamnosus ATCC 53103 and Lactobacillus reuteri DSM 29063, 5x10^9 CFU and 1x10^8 CFU, respectively, per seven drops.
  Flostrum Baby - in children below 12 years of age, 7 drops, twice daily; in children older than 12 years, 14 drops, twice daily.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus ATCC 53103 & Lactobacillus reuteri DSM 29063
- Dicoflor (Active Comparator): The control product will be Dicoflor, which is a food supplement containing L rhamnosus ATCC 53103, 5x10^9 CFU, per five drops.
  Dicoflor - the manufacturer recommends 5-10 drops daily, with no age specification. For the purposes of this study, 5 drops, twice daily, in children below 12 years of age; 10 drops, twice daily, in children older than 12 years.
  Interventions: Dietary Supplement: L rhamnosus ATCC 53103

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus ATCC 53103 & Lactobacillus reuteri DSM 29063 — 7 drops contain Lactobacillus rhamnosus GG 5x10^9 CFU; and Lactobacillus reuteri 1x10^8 CFU.
  Other Names: Flostrum Baby
  Arms: Flostrum Baby
Dietary Supplement: L rhamnosus ATCC 53103 — 5 drops contain Lactobacillus rhamnosus 5x10^9 CFU.
  Other Names: Dicoflor
  Arms: Dicoflor

SUMMARY:
This study will use a noninferiority design to examine whether the administration of L rhamnosus ATCC 53103 &amp;amp;amp;amp;amp;amp; L reuteri DSM 29063 (Flostrum Baby) is no worse than (or as good as) the administration of a recommended probiotic L rhamnosus ATCC 53103 (commercially available as Dicoflor, hereafter a reference product) for the prevention of antibiotic-associated diarrhea in children,

DETAILED DESCRIPTION:
The recruitment will take place in hospitalized patients at the Pediatric Department of St. Hedwig of Silesia Hospital, Trzebnica, Poland. Additionally, patients treated at the out-patient clinics collaborating with the St. Hedwig of Silesia Hospital will be recruited. The involvement of other recruiting wards and/or sites are under consideration provided that the personnel are adequately trained and competent in conducting clinical trials. The start of the recruitment is planned in March 2020 and should be completed within the following 2 years.

The test product will be Flostrum Baby, which is a food supplement consisting of two bacterial strains: Lactobacillus rhamnosus ATCC 53103 and Lactobacillus reuteri DSM 29063, 5x10^9 CFU and 1x10^8 CFU, respectively, per seven drops.

The control product will be Dicoflor, which is a food supplement containing L rhamnosus ATCC 53103, 5x10^9 CFU, per five drops.

Caregivers will receive oral and written information regarding the study. Written informed consent will be obtained by the physicians involved in the study. Participants will be randomized within 24 hours after the initiation of the antibiotic administration.

Throughout the study period, healthcare providers and/or caregivers will record the number and consistency of stools in a standard stool diary. To record stool consistency, in children younger than 1 year, the Amsterdam Infant Stool Scale (AISS)9 will be used, and loose or watery stools will correspond to A-consistency. In children older than 1 year, the Bristol Stool Form (BSF) scale10 will be used, and loose or watery stools will correspond to scores of 5- 7. In the case of missing or incomplete data, data from hospital charts will be obtained. At any time, caregivers will have the right to withdraw the participating child from the study; they will be not obliged to give reasons for this decision, and there will be no effect on subsequent physician and/or institutional medical care.

In the event of loose or watery stools, the presence of viral or bacterial pathogens in the stool samples will be investigated. The presence of viral pathogens will be checked by using a standard rapid, qualitative, chromatographic immunoassay that simultaneously detects rotaviruses, adenoviruses, and noroviruses. Standard microbiological techniques will be used to isolate and identify bacterial pathogens (Salmonella spp, Shigella spp, Campylobacter spp, and Yersinia spp). C. difficile toxins A and B will be identified by standard enzyme immunoassay.

All study participants will be followed up for the duration of the intervention (antibiotic treatment) and then for up to 1 week after the intervention.

ELIGIBILITY:
Inclusion criteria:

1. age younger than 18 years;
2. oral or intravenous antibiotic therapy which started within 24 hours of enrolment;
3. signed informed consent.

Exclusion criteria:

1. pre-existing acute or chronic diarrhea, history of chronic gastrointestinal disease (e.g. inflammatory bowel disease, cystic fibrosis, coeliac disease, food allergy) or other severe chronic diseases (eg, neoplastic diseases),
2. major medical problems (eg. immunocompromised, major developmental or genetic abnormality);
3. taking any of the study products (or probiotic strains included in the study products) at the time of study commencement;
4. use of antibiotics within 4 weeks prior to enrolment,
5. prematurity;
6. exclusive breastfeeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 892 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Antibiotic-associated diarrhea (3 or more loose or watery stools (a score of A on the AIS Scale or 5-7 on the BSF scale) per day in a 24-hour period, caused by C. difficile infection or of otherwise unexpla | From the date of randomisation up to 7th day after antibiotic cessation

SECONDARY OUTCOMES:
• Any diarrhea (defined as ≥ 3 loose or watery stools per day for a minimum of 24 hours regardless of its etiology). | From the date of randomisation up to 7th day after antibiotic cessation
• C difficile-associated diarrhea (CDAD) (diarrhea defined as above caused by C. difficile confirmed by the presence of toxin-producing C. difficile in stools (positive toxin tests)) | From the date of randomisation up to 7th day after antibiotic cessation
• The duration of diarrhea (defined as the time until the normalization of stool consistency according to the BSF or AISS scale (on BSF scale, numbers 1, 2, 3 and 4; on AISS scale, letters B or C), and the presence of normal stools for 48 hours). | From the date of randomisation up to 7th day after antibiotic cessation
• Discontinuation of the antibiotic treatment due to severity of diarrhea. | From the date of randomisation up to 7th day after antibiotic cessation
• Hospitalization caused by diarrhea in outpatient | From the date of randomisation up to 7th day after antibiotic cessation
• Adverse events. | From the date of randomisation up to 7th day after antibiotic cessation
Number and consistency of stools | From the date of randomisation up to 7th day after antibiotic cessation

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Szajewska, MD, Study Chair — The Medical Univ of Warsaw, Dept of Paediatrics; Henryk Szymański, MD, Principal Investigator — Pediatric Department of St. Hedwig of Silesia Hospital
Locations (1):
- Department of Paediatrics, St. Hedwig of Silesia Hospital, Trzebnica, Poland

IPD SHARING:
Plan to Share IPD: No